CLINICAL TRIAL: NCT05612503
Title: Virtual Reality-based Exercises' Effects on Pulmonary Functions, Cardiopulmonary Capacity, Functional Performance, and Quality of Life in Children With Repaired Congenital Diaphragmatic Hernia
Brief Title: Virtual Reality and Congenital Diaphragmatic Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/2021/0074
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Virtual Reality; Congenital Diaphragmatic Hernia; Children
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy program (Sham Comparator): For 15 minutes, each child in both groups perform the following specific respiratory exercises: resistance-based diaphragm strengthening exercises, breathing exercises.
  Interventions: Other: Traditional physical therapy program
- Virtual reality-based exercises (Experimental): Following a session of traditional physical therapy, the children in study group toke 30 minutes rest then they joined in a 30-minute VR exercise session using Nintendo Wii systems.
  Interventions: Other: Traditional physical therapy program; Other: Virtual reality-based exercises

INTERVENTIONS:
Other: Traditional physical therapy program — resistance-based diaphragm strengthening exercises, breathing exercises to increase costal or chest breathing, and breathing exercises to relax the breathing muscles.
Other: Virtual reality-based exercises — Virtual reality exercise using Nintendo Wii systems. As game interfaces, the Nintendo Wii systems employ haptic sensor-based controllers and a balance board.
  Arms: Virtual reality-based exercises

SUMMARY:
The study has been designed to investigate the effect of 12 weeks of using virtual reality based exercises on pulmonary functions, exercise capacity, functional performance, and quality of life in children with surgically-repaired congenital diaphragmatic hernia.

DETAILED DESCRIPTION:
Children with CDH have significant disruptions in their quality of life (QoL) due to their poor health, in this randomized controlled clinical trial, one important aspect of virtual reality is the interactivity of children and their interests in choosing the exercised game. Each child in two groups perform a specific virtual reality based respiratory exercises for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 10 years.
* BMI was between 20 and 24 kg/m2.
* surgically-repaired congenital diaphragmatic hernia.
* respiratory distress symptoms.
* under follow-up care in pediatric and physical therapy clinic.

Exclusion Criteria:

* Children were excluded if they have growth abnormality.
* neuromotor disorders.
* children with cardiac problems.
* unable to do understand all procedures.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test, forced expiratory volume in the first second | From date of randomization (first week of intervention)
  A pulmonary function test was conducted for all participants using a spirometry analyzer (Autospiro-507; Minato Medical Science; Osaka. Japan).
Pulmonary function test, forced expiratory volume in the first second | after 12 weeks
  A pulmonary function test was conducted for all participants using a spirometry analyzer (Autospiro-507; Minato Medical Science; Osaka. Japan).
Pulmonary function test, forced vital capacity | From date of randomization (first week of intervention)
  A pulmonary function test was conducted for all participants using a spirometry analyzer (Autospiro-507; Minato Medical Science; Osaka. Japan).
Pulmonary function test, forced vital capacity | after 12 weeks
  A pulmonary function test was conducted for all participants using a spirometry analyzer (Autospiro-507; Minato Medical Science; Osaka. Japan).
Pulmonary function test, FEV1/FVC ratio | From date of randomization (first week of intervention)
  performed using a spirometer (Autospiro-507; Minato Medical Science; Osaka. Japan)., (forced expiratory volume in the first second/ forced vital capacity) FEV1/FVC ratio was recorded.
Pulmonary function test, FEV1/FVC ratio | after 12 weeks
  performed using a spirometer (Autospiro-507; Minato Medical Science; Osaka. Japan)., (forced expiratory volume in the first second/ forced vital capacity) FEV1/FVC ratio was recorded.
Exercise capacity assessment | From date of randomization (first week of intervention)
  Cardiopulmonary pulmonary exercise test using the Bruce treadmill test was used to asess the exercise capacity.
Exercise capacity assessment | after 12 weeks
  Cardiopulmonary pulmonary exercise test using the Bruce treadmill test was used to asess the exercise capacity.

SECONDARY OUTCOMES:
Functional performance assessment | From date of randomization (first week of intervention)
  Functional performance was assessed through using the 6-min walk test.
Functional performance assessment | after 12 weeks
  Functional performance was assessed through using the 6-min walk test.
Pediatric Quality of Life Inventory | From date of randomization (first week of intervention)
  Quality of life was evaluated using self-report Pediatric Quality of Life Inventory (PedsQL), it is multidimensional measures of HRQL in children and adolescents, it includes 23 items distributed among 4 domains [physical (8 items) , emotional( 5 items), social ( 5 items ), and school functions ( 3 items )] including 23 items. It provides child self-report and parents report with 5- points scale ( 0 means never, and 4 means almost always).
Pediatric Quality of Life Inventory | after 12 weeks
  Quality of life was evaluated using self-report Pediatric Quality of Life Inventory (PedsQL), it is multidimensional measures of HRQL in children and adolescents, it includes 23 items distributed among 4 domains [physical (8 items) , emotional( 5 items), social ( 5 items ), and school functions ( 3 items )] including 23 items. It provides child self-report and parents report with 5- points scale ( 0 means never, and 4 means almost always).

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Study Director — Prince Sattam Bin Abdulaziz University; Ragab Elnaggar,, PhD, Study Chair — Prince Sattam Bin Abdulaziz University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] van den Hout L, Schaible T, Cohen-Overbeek TE, Hop W, Siemer J, van de Ven K, Wessel L, Tibboel D, Reiss I. Actual outcome in infants with congenital diaphragmatic hernia: the role of a standardized postnatal treatment protocol. Fetal Diagn Ther. 2011;29(1):55-63. doi: 10.1159/000322694. Epub 2011 Feb 3. PMID 21325859
- [Result] Zaccara A, Turchetta A, Calzolari A, Iacobelli B, Nahom A, Lucchetti MC, Bagolan P, Rivosecchi M, Coran AG. Maximal oxygen consumption and stress performance in children operated on for congenital diaphragmatic hernia. J Pediatr Surg. 1996 Aug;31(8):1092-4; discussion 1095. doi: 10.1016/s0022-3468(96)90094-9. PMID 8863241
- [Result] Rutkowski S, Szczegielniak J, Szczepanska-Gieracha J. Evaluation of the Efficacy of Immersive Virtual Reality Therapy as a Method Supporting Pulmonary Rehabilitation: A Randomized Controlled Trial. J Clin Med. 2021 Jan 18;10(2):352. doi: 10.3390/jcm10020352. PMID 33477733